CLINICAL TRIAL: NCT06604767
Title: A Phase 1, Dose-Escalation, Randomized, Active-Controlled, Modified Double-Blind, Parallel-Group, Multi-Arm Study to Investigate the Safety and Immunogenicity of a Combined Respiratory Syncytial Virus/Human Metapneumovirus/Parainfluenza Virus Type 3 Vaccine Candidate in Adult Participants Aged 60 Years and Older
Brief Title: Study of a Respiratory Syncytial Virus/Human Metapneumovirus/Parainfluenza Virus Type 3 Vaccine Candidate in Adults Aged 60 Years and Older
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VBD00006; U1111-1304-9362 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus Infection; Metapneumovirus Infection; Parainfluenzae Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Paramyxoviridae Infections

STUDY DESIGN:
Intervention Model Description: Modified double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: -Investigators, Sponsor and study site staff, laboratory personnel, and participants will be blinded. Study staff preparing/administering the study interventions will be unblinded. Specific Sponsor personnel will be unblinded for the assessment of safety in the sentinel cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- PIV3 Dose 1 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: parainfluenza virus type 3 vaccine (PIV3)
- PIV3 Dose 2 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: parainfluenza virus type 3 vaccine (PIV3)
- PIV3 Dose 3 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: parainfluenza virus type 3 vaccine (PIV3)
- PIV3 Dose 4 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: parainfluenza virus type 3 vaccine (PIV3)
- RSV/hMPV /PIV3 Formulation 1 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: RSV/hMPV/PIV3 vaccine
- RSV/hMPV Formulation 1 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: RSV/hMPV vaccine
- RSV/hMPV Formulation 2 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: RSV/hMPV vaccine
- RSV vaccine 1 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: RSV vaccine 1
- RSV vaccine 2 (Experimental): Participants will receive a single intramuscular (IM) injection at Day 1
  Interventions: Biological: RSV vaccine 2

INTERVENTIONS:
Biological: parainfluenza virus type 3 vaccine (PIV3) — Pharmaceutical form:Frozen liquid solution -Route of administration:Intramuscular
  Arms: PIV3 Dose 1; PIV3 Dose 2; PIV3 Dose 3; PIV3 Dose 4
Biological: RSV/hMPV/PIV3 vaccine — Pharmaceutical form:Frozen liquid solution-Route of administration:Intramuscular
  Arms: RSV/hMPV /PIV3 Formulation 1
Biological: RSV/hMPV vaccine — Pharmaceutical form:Frozen liquid solution-Route of administration:Intramuscular
  Arms: RSV/hMPV Formulation 1; RSV/hMPV Formulation 2
Biological: RSV vaccine 1 — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Arms: RSV vaccine 1
Biological: RSV vaccine 2 — Pharmaceutical form:Frozen liquid solution-Route of administration:Intramuscular
  Arms: RSV vaccine 2

SUMMARY:
The purpose of this phase 1 study is to evaluate whether the vaccine is safe and can help the body to develop germ fighting agents called "antibodies" (immunogenicity) against the respiratory syncytial virus (RSV), human metapneumovirus (hMPV), and parainfluenza virus type 3 (PIV3). The study will use different doses of PIV3 only and different combinations of RSV/hMPV/PIV3 or RSV/hMPV or only RSV vaccine in adults aged 60 years and older.

DETAILED DESCRIPTION:
The study duration will be up to approximately 12 months minus the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older on the day of inclusion (means from the means from the day of the 60th birthday).
* Informed consent form (ICF) has been signed and dated
* A female participant is eligible to participate if she is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

-Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Presence of unsolicited systemic adverse events (AEs) reported in the 30 minutes after each vaccination | Within 30 minutes after each vaccination
  Number of participants experiencing immediate unsolicited systemic AEs
Presence of solicited administration site reactions within 7 days after vaccination | Within 7 days after vaccination
  Number of participants reporting:
  - injection site reactions: pain, erythema and swelling
Presence of solicited systemic reactions within 7 days after vaccination | Within 7 days after vaccination
  Number of participants reporting:
  * systemic reactions: fever, headache, fatigue, myalgia, arthralgia and chills
Presence of unsolicited AEs within 28 days after vaccination | Within 28 days after vaccination
  Number of participants experiencing unsolicited AEs
Presence of serious adverse events (SAEs) | Within 6 months after vaccination
  Number of participants experiencing SAEs regardless of causality
Presence of adverse events of special interest (AESIs) | Within 6 months after vaccination
  Number of participants experiencing AESIs regardless of causality
Presence of related SAEs throughout the study | Throughout the study, approximately 12 months
  Number of participants experiencing related SAEs regardless of causality
Presence of related AESIs throughout the study | Throughout the study, approximately 12 months
  Number of participants experiencing related AESIs regardless of causality
Presence of related fatal SAEs throughout the study | Throughout the study, approximately 12 months
  Number of participants experiencing related fatal SAEs regardless of causality
Presence of out-of-range biological test results (including shift from baseline values) | Within 7 days after vaccination
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test, including shift from baseline values)

SECONDARY OUTCOMES:
RSV A serum neutralizing antibody (nAb) titers at pre-vaccination (Day 01) and post-vaccination (Day 29) in the RSV/hMPV +/- PIV3 and RSV vaccines | At Day 01 and Day 29
  Antibody titers are expressed as GMTs at pre-vaccination and post-vaccination
RSV B serum nAb titers at pre-vaccination (Day 01) and post-vaccination (Day 29) in the RSV/hMPV +/- PIV3 and RSV vaccines | At Day 01 and Day 29
  Antibody titers are expressed as GMTs at pre-vaccination and post-vaccination
hMPV A serum nAb titers at pre-vaccination (Day 01) and post-vaccination (Day 29) in the RSV/hMPV +/- PIV3 vaccines | At Day 01 and Day 29
  Antibody titers are expressed as GMTs at pre-vaccination and post-vaccination
PIV3 serum nAb titers at pre-vaccination (Day 01) and post-vaccination (Day 29) in the RSV/hMPV/PIV3 and PIV3 vaccines | At Day 01 and Day 29
  Antibody titers are expressed as GMTs at pre-vaccination and post-vaccination

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (8):
  - Investigational Site Number : 0360006, Blacktown, New South Wales
  - Investigational Site Number : 0360001, Botany, New South Wales
  - Investigational Site Number : 0360009, Brookvale, New South Wales
  - Investigational Site Number : 0360005, Kanwal, New South Wales
  - Investigational Site Number : 0360004, Miranda, New South Wales
  - Investigational Site Number : 0360008, Herston, Queensland
  - Investigational Site Number : 0360003, Bayswater, Victoria
  - Investigational Site Number : 0360002, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBD00006 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26144&tenant=MT_SNY_9011